CLINICAL TRIAL: NCT07365319
Title: A Global, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2/3 Study of EIK1001 in Combination With Pembrolizumab and Chemotherapy in Participants With Stage 4 Non-Small Cell Lung Cancer (TeLuRide-008).
Brief Title: A Safety and Efficacy Study of EIK1001 in Combination With Pembrolizumab and Chemotherapy in Participants With Stage 4 Non-Small Cell Lung Cancer.
Acronym: TeLuRide-008
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eikon Therapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIK1001-008; 2025-525013-23-00 (EU CTIS Number); KEYNOTE-G57 (Other: Merck Sharp & Dohme LLC); MK-3475-G57 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2026-01-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Non Small Cell Lung Cancer (Squamous or Non Squamous); Stage 4 NSCLC
Keywords: Non Small Cell Lung Cancer; EIK1001
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; CP protocol; 130-nm albumin-bound paclitaxel; Carboplatin; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Placebo in Combination with SOC) (Placebo Comparator): Participants in this arm will receive EIK1001 Placebo + Standard of Care (SOC).
  Interventions: Drug: Pembrolizumab (KEYTRUDA®); Drug: Placebo; Drug: Paclitaxel + Carboplatin; Drug: Nab-paclitaxel + Carboplatin; Drug: Pemetrexed + Cisplatin /Carboplatin
- Arm 2 (EIK1001 in Combination with SOC) (Experimental): Participants in this arm will receive EIK1001 (Selected Dose 1) + Standard of Care (SOC).
  Interventions: Drug: EIK1001; Drug: Pembrolizumab (KEYTRUDA®); Drug: Paclitaxel + Carboplatin; Drug: Nab-paclitaxel + Carboplatin; Drug: Pemetrexed + Cisplatin /Carboplatin
- Arm 3 (EIK1001 in Combination with SOC) (Experimental): Participants in this arm will receive EIK1001 (Selected Dose 2) + Standard of Care (SOC).
  Interventions: Drug: EIK1001; Drug: Pembrolizumab (KEYTRUDA®); Drug: Paclitaxel + Carboplatin; Drug: Nab-paclitaxel + Carboplatin; Drug: Pemetrexed + Cisplatin /Carboplatin

INTERVENTIONS:
Drug: EIK1001 — EIK1001 is a Toll like receptor 7/8 (TLR 7/8) dual agonist
  Arms: Arm 2 (EIK1001 in Combination with SOC); Arm 3 (EIK1001 in Combination with SOC)
Drug: Pembrolizumab (KEYTRUDA®) — PD-1 inhibitor
Drug: Placebo — Placebo control
  Arms: Arm 1 (Placebo in Combination with SOC)
Drug: Paclitaxel + Carboplatin — SOC Chemotherapy for squamous NSCLC
Drug: Nab-paclitaxel + Carboplatin — SOC Chemotherapy for squamous NSCLC
Drug: Pemetrexed + Cisplatin /Carboplatin — SOC Chemotherapy for non-squamous NSCLC

SUMMARY:
This is a study to evaluate the safety and efficacy of EIK1001 administered intravenously in combination with pembrolizumab and histologically appropriate chemotherapy for patients with stage 4 NSCLC.

DETAILED DESCRIPTION:
This is a global, multicenter, double-blind, placebo-controlled, randomized adaptive Phase 2/3 study to evaluate the clinical activity and safety of EIK1001 administered IV in combination with pembrolizumab and histologically appropriate chemotherapy (pemetrexed plus either carboplatin or cisplatin) to participants with Stage 4 non-squamous or (carboplatin plus either paclitaxel or nab-paclitaxel) for participants with squamous NSCLC who have not received prior systemic therapy. The study is conducted in 2 phases (Phase 2 and Phase 3) and analyzed in 3 parts (dose optimization, dose expansion and confirmatory hypothesis testing).

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant must be ≥ 18 years old at the time of signing the informed consent.
2. Participant has a life expectancy of at least 3 months.
3. Participant has histologically or cytologically confirmed Stage 4 NSCLC predominately squamous or non-squamous) and is considered a candidate for standard therapy with pembrolizumab and chemotherapy. Participants with NSCLC-NOS (not otherwise specified) will be considered as non-squamous NSCLC.
4. Participant must have documented evidence that mutation-directed therapy is not indicated, based on the absence of tumor-activating mutations or fusions (e.g., but not limited to EGFR, ALK, RET, ROS1, BRAF) for which approved first-line targeted therapies are available to the participant in their respective country.
5. Participant has at least 1 lesion with measurable disease at Baseline according to RECIST 1.1 as determined locally. Lesions situated in a previously irradiated area are considered measurable if progression has been shown in such lesions.
6. Participant has not received prior systemic therapy for advanced/metastatic NSCLC.

   Note: Participants who received adjuvant or neoadjuvant treatment (after surgery and/or radiation therapy) and developed recurrent or metastatic disease more than 1 year after completing therapy are eligible.
7. Participant has an ECOG Performance Status of 0 to 1 assessed no more than 10 days before start of the treatment.
8. Participant has tumor tissue available for PD-L1 testing from a site that was not radiated prior to biopsy, and was obtained, ideally, after diagnosis of metastatic disease. Biopsies obtained prior to receipt of adjuvant/neoadjuvant chemotherapy will be permitted if recent biopsy is not feasible (provided the specimen is < 3yrs old).

Key Exclusion Criteria:

1. has small cell elements present histologically and/or the tumors are not predominantly non-squamous or squamous NSCLC.
2. is currently actively enrolled in or has recently participated in a study of an investigational agent and received investigational therapy within 4 weeks or 5 half-lives (whichever is longer) of administration of EIK1001 or placebo.
3. has had major surgery (< 3 weeks prior to the first dose of study intervention administration).
4. has received a live-virus vaccination within 30 days of the start of study intervention initiation.
5. has received radiation therapy within 7 days of the first dose of study intervention administration.
6. has completed palliative radiotherapy within 7 days of the first dose of study intervention administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2026-05-18 (Estimated); Primary Completion 2035-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Through study completion, up to 6 years
  Progression-free survival (PFS) is defined as the time from the first dose of the study medication to the first documented disease progression according to RECIST 1.1 by BICR, or death due to any cause, whichever occurs first
Overall survival (OS) | Through study completion, up to 10 years
  OS defined as the time from the first dose of study medication to death due to any cause
Objective Response (OR) | Through study completion, up to 6 years
  Objective response (OR) is defined as participants who demonstrate complete response (CR) or partial response (PR) by RECIST 1.1 as assessed by the Investigator, adverse events (AEs), and discontinuation of study intervention due to an AE (Dose Optimization Only).

SECONDARY OUTCOMES:
Objective response (OR) | Up to 6 years
  Objective response (OR) is defined as participants who have a confirmed complete response (CR) or partial response (PR) according to RECIST 1.1 by BICR
Duration of response (DOR) | Up to 6 years
  DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first, in participants demonstrating CR or PR, according to RECIST 1.1 by BICR.
Progression-free survival (PFS) by Investigator | Up to 6 years
  Progression-free survival (PFS) is defined as the time from the first dose of the study medication to the first documented disease progression according to RECIST 1.1 by Investigator, or death due to any cause, whichever occurs first.
Overall Response Rate (ORR) by Investigator | Up to 6 years
  Objective Response as defined by participants who demonstrate confirmed CR or PR according to RECIST 1.1 by Investigator.
Duration of Response (DOR) by Investigator | Up to 6 years
  DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first, in participants demonstrating CR or PR, according to RECIST 1.1 by Investigator.
Incidence of Adverse Events (AEs) | Up to 2.5 years
  Adverse Events (AEs) and discontinuation of study treatment due to any AE.

CONTACTS AND LOCATIONS:
Overall Officials: Etah Kurland, MD, Study Director — Eikon Therapeutics

IPD SHARING:
Plan to Share IPD: No